CLINICAL TRIAL: NCT01106677
Title: A Randomized, Double-Blind, Placebo and Active-Controlled, 4-Arm, Parallel Group, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Canagliflozin in the Treatment of Subjects With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin Monotherapy
Brief Title: The CANTATA-D Trial (CANagliflozin Treatment and Trial Analysis - DPP-4 Inhibitor Comparator Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017023; 28431754DIA3006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-04-01; First posted 2010-04-20 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes mellitus; Canagliflozin; Placebo; Sitagliptin; Januvia; Metformin Immediate Release (IR); Hemoglobin A1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin; Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Canagliflozin 100 mg (Experimental): Each patient will receive 100 mg of canagliflozin once daily for 52 weeks with protocol-specified doses of metformin immediate release.
  Interventions: Drug: Canagliflozin; Drug: Metformin immediate release
- Canagliflozin 300 mg (Experimental): Each patient will receive 300 mg of canagliflozin once daily for 52 weeks with protocol-specified doses of metformin immediate release.
  Interventions: Drug: Canagliflozin; Drug: Metformin immediate release
- Sitagliptin 100 mg (Active Comparator): Each patient will receive 100 mg of sitagliptin once daily for 52 weeks with protocol-specified doses of metformin immediate release.
  Interventions: Drug: Sitagliptin; Drug: Metformin immediate release
- Placebo/Sitagliptin (Other): Each patient will receive matching placebo once daily for 26 weeks and will then switch from placebo to 100 mg of sitagliptin once daily until Week 52. Placebo and sitagliptin will be given with protocol-specified doses of metformin immediate release.
  Interventions: Drug: Placebo; Drug: Sitagliptin; Drug: Metformin immediate release

INTERVENTIONS:
Drug: Placebo — One matching placebo capsule orally (by mouth) once daily for 26 weeks with protocol-specified doses of metformin immediate release.
  Arms: Placebo/Sitagliptin
Drug: Canagliflozin — One 100 mg or 300 mg over-encapsulated tablet orally once daily for 52 weeks with protocol-specified doses of metformin immediate release.
  Arms: Canagliflozin 100 mg; Canagliflozin 300 mg
Drug: Sitagliptin — One 100 mg over-encapsulated tablet orally once daily for 52 weeks (sitagliptin 100 mg arm) or once daily beginning at Week 26 until Week 52 (placebo/sitagliptin arm). Sitagliptin will be given with protocol-specified doses of metformin immediate release.
  Arms: Placebo/Sitagliptin; Sitagliptin 100 mg
Drug: Metformin immediate release — The patient's stable dose of metformin immediate release background therapy should be continued throughout the study.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of canagliflozin compared with sitagliptin and placebo in patients with type 2 diabetes mellitus who are receiving treatment with metformin monotherapy (i.e., treatment with a single drug) and have inadequate glycemic (blood sugar) control.

DETAILED DESCRIPTION:
Canagliflozin is a drug that is being tested to see if it may be useful in treating patients diagnosed with type 2 diabetes mellitus (T2DM). This is a randomized (study drug assigned by chance), double-blind (neither the patient nor the study doctor will know the identity of assigned study drug), placebo- and active-controlled, parallel-group, 4-arm (4 treatment groups) multicenter study to determine the efficacy, safety, and tolerability of canagliflozin (100 mg and 300 mg) compared to placebo (a capsule that looks like all the other treatments but has no real medicine) and an active-control (sitagliptin 100 mg, an antihyperglycemic agent) in patients with T2DM who are not achieving an adequate response from current antihyperglycemic therapy with metformin Immediate Release (IR) to control their diabetes. Approximately 1,260 patients with T2DM who are receiving treatment with metformin IR and have inadequate glycemic (blood sugar) will receive once-daily treatment with canagliflozin (100 mg or 300 mg), sitagliptin 100 mg, or placebo capsules for 26 weeks (Period I) followed by another 26-weeks where patients treated with canagliflozin (100 mg or 300 mg) or sitagliptin 100 mg will continue treatment for an additional 26 weeks and patients treated with placebo will be switched to active double-blind treatment with sitagliptin 100 mg capsules administered once-daily for 26 weeks (Period II). In addition, all patients will take protocol specified stable doses of metformin IR along with assigned study drug for the duration of the study. Patients will participate in the study for approximately 59 to 71 weeks. During the study, if a patient's fasting blood sugar remains high despite treatment with study drug, metformin IR, and reinforcement with diet and exercise, the patient will receive treatment with glimepiride (rescue therapy) consistent with local prescribing information. During treatment, patients will be monitored for safety by review of adverse events, results from laboratory tests, 12-lead electrocardiograms (ECGs), vital sign measurements, body weight, physical examinations, and self-monitored blood glucose (SMGB) measurements. The primary outcome measure in the study is to assess the effect of canagliflozin relative to placebo on hemoglobin A1c (HbA1c) after 26 weeks of treatment. Study drug will be taken orally (by mouth) once daily before the first meal each day unless otherwise specified. Patients will take single-blind placebo for 2 weeks before randomization. After randomization, patients in the study will take double-blind canagliflozin (100 mg or 300 mg) or sitagliptin 100 mg for 52 weeks OR placebo for 26 weeks switched to double-blind treatment with sitaliptin 100 mg for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of T2DM and be currently treated with metformin IR
* Patients in the study must have a HbA1c between >=7 and <=10.5%
* Patients must have a fasting plasma glucose (FPG) <270 mg/dL (15 mmol/L)

Exclusion Criteria:

* History of diabetic ketoacidosis, type 1 diabetes mellitus (T1DM), pancreas or beta cell transplantation, diabetes secondary to pancreatitis or pancreatectomy, or a severe hypoglycemic episode within 6 months before screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1284 (Actual)
Dates: Start 2010-05; Primary Completion 2011-10 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (125):
- United States (45):
  - Little Rock, Arkansas
  - Fountain Valley, California
  - National City, California
  - Northridge, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Bradenton, Florida
  - Brooksville, Florida
  - DeFuniak Springs, Florida
  - Hialeah, Florida
  - Niceville, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Champaign, Illinois
  - Avon, Indiana
  - Fishers, Indiana
  - Franklin, Indiana
  - West Des Moines, Iowa
  - Wichita, Kansas
  - Munfordville, Kentucky
  - Portland, Maine
  - Benzonia, Michigan
  - Interlochen, Michigan
  - Troy, Michigan
  - Picayune, Mississippi
  - Florissant, Missouri
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Mansfield, New Jersey
  - New Hyde Park, New York
  - Asheboro, North Carolina
  - Charlotte, North Carolina
  - Kettering, Ohio
  - Oregon City, Oregon
  - Altoona, Pennsylvania
  - Tipton, Pennsylvania
  - East Providence, Rhode Island
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Nashville, Tennessee
  - New Braunfels, Texas
  - San Antonio, Texas
  - Bountiful, Utah
  - Spokane, Washington
- Argentina (3):
  - Buenos Aires
  - Mendoza
  - San Juan
- Bulgaria (4):
  - Pleven
  - Plovdiv
  - Sevlievo
  - Sofia
- Colombia (3):
  - Barranquilla
  - Bogotá
  - Medellín
- Czechia (5):
  - Beroun
  - Pardubice
  - Pilsen
  - Rychnov nad Kněžnou
  - Tábor
- Tallinn, Estonia
- Greece (2):
  - Piraeus
  - Thessalonikis
- India (10):
  - Ahmedabad, Gujarat
  - Aurangabad
  - Bangalore
  - Bangalore, Karnataka
  - Belagavi
  - Coimbatore
  - Mumbai
  - Nagpur
  - Pune
  - Trivandrum
- Latvia (4):
  - Daugavpils
  - Limbaži
  - Riga
  - Talsi
- Malaysia (4):
  - Kelantan
  - Kuala Lumpur
  - Kuala Selangor
  - Pulau Pinang
- Mexico (5):
  - Culiacán
  - Guadalajara
  - Monterrey
  - Querétaro
  - Tampico
- Lima 1 Lima Lima, Peru
- Poland (5):
  - Lodz
  - Lublin
  - Wroclaw
  - Zgierz
  - Łęczyca
- Portugal (4):
  - Aveiro
  - Leiria
  - Lisbon
  - Portalegre
- San Juan, Puerto Rico
- Russia (6):
  - Chelyabinsk
  - Dzerzhinsky Moscow Region
  - Kemerovo
  - Penza
  - Saint Petersburg
  - Yekaterinburg
- Singapore, Singapore
- Slovakia (5):
  - Banská Bystrica
  - Bratislava
  - Košice
  - Šahy
  - Trebišov
- Sweden (2):
  - Gothenburg
  - Stockholm
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
- Turkey (Türkiye) (5):
  - Ankara
  - Antalya
  - Istanbul
  - Izmir
  - Konya
- Ukraine (6):
  - Donetsk
  - Ivano-Frankivsk
  - Kiev
  - Sumy
  - Vinnitsa
  - Zaporizhzhya

REFERENCES:
- [Derived] Cai J, Delahanty LM, Akapame S, Slee A, Traina S. Impact of Canagliflozin Treatment on Health-Related Quality of Life among People with Type 2 Diabetes Mellitus: A Pooled Analysis of Patient-Reported Outcomes from Randomized Controlled Trials. Patient. 2018 Jun;11(3):341-352. doi: 10.1007/s40271-017-0290-4. PMID 29313267
- [Derived] Davies MJ, Merton K, Vijapurkar U, Yee J, Qiu R. Efficacy and safety of canagliflozin in patients with type 2 diabetes based on history of cardiovascular disease or cardiovascular risk factors: a post hoc analysis of pooled data. Cardiovasc Diabetol. 2017 Mar 21;16(1):40. doi: 10.1186/s12933-017-0517-7. PMID 28327140
- [Derived] Pfeifer M, Townsend RR, Davies MJ, Vijapurkar U, Ren J. Effects of canagliflozin, a sodium glucose co-transporter 2 inhibitor, on blood pressure and markers of arterial stiffness in patients with type 2 diabetes mellitus: a post hoc analysis. Cardiovasc Diabetol. 2017 Feb 27;16(1):29. doi: 10.1186/s12933-017-0511-0. PMID 28241822
- [Derived] Gilbert RE, Mende C, Vijapurkar U, Sha S, Davies MJ, Desai M. Effects of Canagliflozin on Serum Magnesium in Patients With Type 2 Diabetes Mellitus: A Post Hoc Analysis of Randomized Controlled Trials. Diabetes Ther. 2017 Apr;8(2):451-458. doi: 10.1007/s13300-017-0232-0. Epub 2017 Feb 14. PMID 28197834
- [Derived] Qiu R, Balis D, Xie J, Davies MJ, Desai M, Meininger G. Longer-term safety and tolerability of canagliflozin in patients with type 2 diabetes: a pooled analysis. Curr Med Res Opin. 2017 Mar;33(3):553-562. doi: 10.1080/03007995.2016.1271780. Epub 2017 Jan 4. PMID 27977934
- [Derived] John M, Cerdas S, Violante R, Deerochanawong C, Hassanein M, Slee A, Canovatchel W, Hamilton G. Efficacy and safety of canagliflozin in patients with type 2 diabetes mellitus living in hot climates. Int J Clin Pract. 2016 Sep;70(9):775-85. doi: 10.1111/ijcp.12868. PMID 27600862
- [Derived] Schernthaner G, Lavalle-Gonzalez FJ, Davidson JA, Jodon H, Vijapurkar U, Qiu R, Canovatchel W. Canagliflozin provides greater attainment of both HbA1c and body weight reduction versus sitagliptin in patients with type 2 diabetes. Postgrad Med. 2016 Nov;128(8):725-730. doi: 10.1080/00325481.2016.1210988. Epub 2016 Jul 26. PMID 27391951
- [Derived] Watts NB, Bilezikian JP, Usiskin K, Edwards R, Desai M, Law G, Meininger G. Effects of Canagliflozin on Fracture Risk in Patients With Type 2 Diabetes Mellitus. J Clin Endocrinol Metab. 2016 Jan;101(1):157-66. doi: 10.1210/jc.2015-3167. Epub 2015 Nov 18. PMID 26580237
- [Derived] Lavalle-Gonzalez FJ, Eliaschewitz FG, Cerdas S, Chacon Mdel P, Tong C, Alba M. Efficacy and safety of canagliflozin in patients with type 2 diabetes mellitus from Latin America. Curr Med Res Opin. 2016;32(3):427-39. doi: 10.1185/03007995.2015.1121865. Epub 2016 Jan 14. PMID 26579834
- [Derived] Blonde L, Woo V, Mathieu C, Yee J, Vijapurkar U, Canovatchel W, Meininger G. Achievement of treatment goals with canagliflozin in patients with type 2 diabetes mellitus: a pooled analysis of randomized controlled trials. Curr Med Res Opin. 2015 Nov;31(11):1993-2000. doi: 10.1185/03007995.2015.1082991. Epub 2015 Sep 28. PMID 26373629
- [Derived] Gavin JR 3rd, Davies MJ, Davies M, Vijapurkar U, Alba M, Meininger G. The efficacy and safety of canagliflozin across racial groups in patients with type 2 diabetes mellitus. Curr Med Res Opin. 2015;31(9):1693-702. doi: 10.1185/03007995.2015.1067192. Epub 2015 Sep 4. PMID 26121561
- [Derived] Cefalu WT, Stenlof K, Leiter LA, Wilding JP, Blonde L, Polidori D, Xie J, Sullivan D, Usiskin K, Canovatchel W, Meininger G. Effects of canagliflozin on body weight and relationship to HbA1c and blood pressure changes in patients with type 2 diabetes. Diabetologia. 2015 Jun;58(6):1183-7. doi: 10.1007/s00125-015-3547-2. Epub 2015 Mar 27. PMID 25813214
- [Derived] Bailey RA, Vijapurkar U, Meininger G, Rupnow MF, Blonde L. Diabetes-Related Composite Quality End Point Attainment: Canagliflozin Versus Sitagliptin Based on a Pooled Analysis of 2 Clinical Trials. Clin Ther. 2015 May 1;37(5):1045-54. doi: 10.1016/j.clinthera.2015.02.020. Epub 2015 Mar 18. PMID 25795432
- [Derived] Weir MR, Januszewicz A, Gilbert RE, Vijapurkar U, Kline I, Fung A, Meininger G. Effect of canagliflozin on blood pressure and adverse events related to osmotic diuresis and reduced intravascular volume in patients with type 2 diabetes mellitus. J Clin Hypertens (Greenwich). 2014 Dec;16(12):875-82. doi: 10.1111/jch.12425. Epub 2014 Oct 20. PMID 25329038
- [Derived] Usiskin K, Kline I, Fung A, Mayer C, Meininger G. Safety and tolerability of canagliflozin in patients with type 2 diabetes mellitus: pooled analysis of phase 3 study results. Postgrad Med. 2014 May;126(3):16-34. doi: 10.3810/pgm.2014.05.2753. PMID 24918789
- [Derived] Weir MR, Kline I, Xie J, Edwards R, Usiskin K. Effect of canagliflozin on serum electrolytes in patients with type 2 diabetes in relation to estimated glomerular filtration rate (eGFR). Curr Med Res Opin. 2014 Sep;30(9):1759-68. doi: 10.1185/03007995.2014.919907. Epub 2014 May 22. PMID 24786834
- [Derived] Sinclair A, Bode B, Harris S, Vijapurkar U, Mayer C, Fung A, Shaw W, Usiskin K, Desai M, Meininger G. Efficacy and safety of canagliflozin compared with placebo in older patients with type 2 diabetes mellitus: a pooled analysis of clinical studies. BMC Endocr Disord. 2014 Apr 18;14:37. doi: 10.1186/1472-6823-14-37. PMID 24742013
- [Derived] Nyirjesy P, Sobel JD, Fung A, Mayer C, Capuano G, Ways K, Usiskin K. Genital mycotic infections with canagliflozin, a sodium glucose co-transporter 2 inhibitor, in patients with type 2 diabetes mellitus: a pooled analysis of clinical studies. Curr Med Res Opin. 2014 Jun;30(6):1109-19. doi: 10.1185/03007995.2014.890925. Epub 2014 Feb 21. PMID 24517339
- [Derived] Lavalle-Gonzalez FJ, Januszewicz A, Davidson J, Tong C, Qiu R, Canovatchel W, Meininger G. Efficacy and safety of canagliflozin compared with placebo and sitagliptin in patients with type 2 diabetes on background metformin monotherapy: a randomised trial. Diabetologia. 2013 Dec;56(12):2582-92. doi: 10.1007/s00125-013-3039-1. Epub 2013 Sep 13. PMID 24026211

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the efficacy and safety of canagliflozin compared with sitagliptin and placebo in patients with type 2 diabetes mellitus with inadequate control despite treatment with metformin. The study was conducted between 07 April 2010 and 17 August 2012 and recruited patients from 169 study centers in 22 countries worldwide.
Pre-assignment Details: 1,284 patients were randomly allocated to the 4 treatment arms. All patients received at least 1 dose of study drug and were included in the modified intent-to-treat (mITT) analysis set (used for the Week 26 and week 52 efficacy analyses). All 1,284 patients were included in the Week 26 and Week 52 safety analysis sets.
Groups:
- Placebo/Sitagliptin: Each patient received matching placebo once daily for 26 weeks and were then switched from placebo to 100 mg of sitagliptin once daily until Week 52. Placebo and sitagliptin were given with protocol-specified doses of metformin immediate release.
- Canagliflozin 100 mg: Each patient received 100 mg of canagliflozin once daily for 52 weeks with protocol-specified doses of metformin immediate release.
- Canagliflozin 300 mg: Each patient received 300 mg of canagliflozin once daily for 52 weeks with protocol-specified doses of metformin immediate release.
- Sitagliptin 100 mg: Each patient received 100 mg of sitagliptin once daily for 52 weeks with protocol-specified doses of metformin immediate release.
Period: Core Period: Baseline to Week 26
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg | Sitagliptin 100 mg
Started | 183 | 368 | 367 | 366
Completed | 155 | 322 | 323 | 319
Not Completed | 28 | 46 | 44 | 47
Not completed — Adverse Event | 7 | 18 | 6 | 8
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 1 | 6 | 3
Not completed — Physician Decision | 2 | 1 | 3 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 3
Not completed — Withdrawal by Subject | 5 | 3 | 15 | 6
Not completed — Creatinine or eGFR withdrawal criteria | 1 | 2 | 2 | 3
Not completed — Noncompliance with study drug | 1 | 3 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 1 | 2 | 0
Not completed — Product quality complaint | 0 | 1 | 1 | 0
Not completed — Other | 8 | 14 | 8 | 23
Not completed — Pregnancy | 0 | 1 | 0 | 0
Period: Extension Period: Week 26 to Week 52
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg | Sitagliptin 100 mg
Started | 153 (2 pts completed core but did not enter ext: protcol violation(1), lost to f/u(1).) | 316 (6 pts completed core but did not enter ext: not specified(5), withdrawal by subject(1).) | 321 (2 pts completed core but did not enter ext: not specified(1), withdrawal by subject(1).) | 313 (6 pts completed core but did not enter ext: not specified(3), physician decision(2), lost to f/u(1).)
Completed | 138 | 298 | 299 | 285
Not Completed | 15 | 18 | 22 | 28
Not completed — Adverse Event | 1 | 1 | 5 | 9
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 2 | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 2 | 2 | 2
Not completed — Physician Decision | 2 | 3 | 2 | 3
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 2 | 1
Not completed — Creatinine or eGFR withdrawal criteria | 2 | 4 | 3 | 2
Not completed — Unable to take rescue therapy | 0 | 0 | 0 | 1
Not completed — Other | 6 | 5 | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg | Sitagliptin 100 mg | Total
Number analyzed (Participants) | 183 | 368 | 367 | 366 | 1284
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 146 | 314 | 309 | 309 | 1078
  >=65 years | 37 | 54 | 58 | 57 | 206
Age Continuous [Mean (Standard Deviation); unit: years] | 55.3 (9.76) | 55.5 (9.38) | 55.3 (9.19) | 55.5 (9.55) | 55.4 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 194 | 202 | 194 | 679
  Male | 94 | 174 | 165 | 172 | 605
Region Enroll [Number; unit: participants]
  ARGENTINA | 8 | 9 | 15 | 11 | 43
  BULGARIA | 4 | 2 | 1 | 3 | 10
  COLOMBIA | 4 | 15 | 8 | 15 | 42
  CZECH REPUBLIC | 7 | 8 | 8 | 7 | 30
  ESTONIA | 6 | 6 | 3 | 5 | 20
  GREECE | 1 | 1 | 3 | 4 | 9
  INDIA | 13 | 28 | 31 | 22 | 94
  ITALY | 2 | 3 | 3 | 1 | 9
  LATVIA | 3 | 7 | 6 | 10 | 26
  MALAYSIA | 9 | 7 | 11 | 7 | 34
  MEXICO | 12 | 20 | 26 | 18 | 76
  PERU | 16 | 36 | 30 | 37 | 119
  POLAND | 1 | 18 | 14 | 10 | 43
  PORTUGAL | 1 | 1 | 0 | 2 | 4
  RUSSIAN FEDERATION | 15 | 34 | 28 | 22 | 99
  SINGAPORE | 3 | 5 | 3 | 3 | 14
  SLOVAKIA | 12 | 16 | 21 | 17 | 66
  SWEDEN | 3 | 3 | 2 | 4 | 12
  THAILAND | 4 | 9 | 11 | 8 | 32
  TURKEY | 1 | 5 | 11 | 9 | 26
  UKRAINE | 8 | 24 | 29 | 30 | 91
  UNITED STATES | 50 | 111 | 103 | 121 | 385

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean change in HbA1c from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin or sitagliptin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: Analysis used mITT analysis set (all randomized patients who received at least 1 dose of study drug). Last-observation-carried-forward method used for missing Week 26 values. Measurements taken pre-rescue used as last observation in patients receiving glycemic rescue therapy. Table includes only patients with both baseline and post baseline values.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 181 | 365 | 360 | 354
Percent | -0.17 (0.060) | -0.79 (0.044) | -0.94 (0.044) | -0.82 (0.044)
Statistical Analysis 1: Comparison: Placebo/Sitagliptin vs Canagliflozin 100 mg; Test type: Non-Inferiority or Equivalence — Power calculation: assuming a difference between canagliflozin and placebo of 0.5% and a common standard deviation of 1.0%, and using a 2-sample, 1-sided t-test with a Type I error rate of 0.05, it was estimated that 86 subjects per group would provide 90% power to demonstrate superiority of canagliflozin over placebo; p < 0.001, ANCOVA; Least-Squares Mean Difference = -0.62, 95% CI 2-sided [-0.758 to -0.481], Standard Error of Mean 0.071
Statistical Analysis 2: Comparison: Placebo/Sitagliptin vs Canagliflozin 300 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA; Least-Squares Mean Difference = -0.77, 95% CI 2-sided [-0.914 to -0.636], Standard Error of Mean 0.071
Statistical Analysis 3: Comparison: Placebo/Sitagliptin vs Sitagliptin 100 mg; Test type: Superiority or Other; ANCOVA — No formal statistical comparison was conducted; Least-Squares Mean Difference = -0.66, 95% CI 2-sided [-0.795 to -0.516], Standard Error of Mean 0.071

2. Secondary Outcome: Percentage of Patients With HbA1c <7% at Week 26
Description: The table below shows the percentage of patients with HbA1c <7% at Week 26 in each treatment group. The statistical analyses show the treatment differences between each canagliflozin or sitagliptin group and placebo.
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 181 | 365 | 360 | 354
Percentage of patients | 29.8 | 45.5 | 57.8 | 54.5
Statistical Analysis 1: Comparison: Placebo/Sitagliptin vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.29, 95% CI 2-sided [1.50 to 3.50]
Statistical Analysis 2: Comparison: Placebo/Sitagliptin vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.39, 95% CI 2-sided [2.85 to 6.77]

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean change in FPG from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin or sitagliptin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 181 | 365 | 360 | 354
mg/dL | 2.47 (2.576) | -27.3 (1.873) | -37.8 (1.893) | -20.2 (1.908)
Statistical Analysis 1: Comparison: Placebo/Sitagliptin vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -29.8, 95% CI 2-sided [-35.76 to -23.81], Standard Error of Mean 3.044
Statistical Analysis 2: Comparison: Placebo/Sitagliptin vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -40.3, 95% CI 2-sided [-46.25 to -34.26], Standard Error of Mean 3.055
Statistical Analysis 3: Comparison: Placebo/Sitagliptin vs Sitagliptin 100 mg; Test type: Superiority or Other; ANCOVA — No formal statistical comparison was conducted; Least-Squares Mean Difference = -22.7, 95% CI 2-sided [-28.70 to -16.69], Standard Error of Mean 3.060

4. Secondary Outcome: Change in 2-hour Post-prandial Glucose From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean change in 2-hour post-prandial glucose from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin or sitagliptin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 129 | 298 | 288 | 295
mg/dL | -9.79 (4.860) | -47.9 (3.305) | -57.1 (3.356) | -49.3 (3.340)
Statistical Analysis 1: Comparison: Placebo/Sitagliptin vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -38.1, 95% CI 2-sided [-49.14 to -27.16], Standard Error of Mean 5.601
Statistical Analysis 2: Comparison: Placebo/Sitagliptin vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -47.3, 95% CI 2-sided [-58.40 to -36.29], Standard Error of Mean 5.635
Statistical Analysis 3: Comparison: Placebo/Sitagliptin vs Sitagliptin 100 mg; Test type: Superiority or Other; ANCOVA — No formal statistical comparison was conducted; Least-Squares Mean Difference = -39.6, 95% CI 2-sided [-50.56 to -28.55], Standard Error of Mean 5.608

5. Secondary Outcome: Percent Change in Body Weight From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean percent change in body weight from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin or sitagliptin group minus placebo) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 181 | 365 | 360 | 355
Percent change | -1.2 (0.3) | -3.7 (0.2) | -4.2 (0.2) | -1.2 (0.2)
Statistical Analysis 1: Comparison: Placebo/Sitagliptin vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -2.5, 95% CI 2-sided [-3.1 to -1.9], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Placebo/Sitagliptin vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -2.9, 95% CI 2-sided [-3.5 to -2.3], Standard Error of Mean 0.3
Statistical Analysis 3: Comparison: Placebo/Sitagliptin vs Sitagliptin 100 mg; Test type: Superiority or Other; ANCOVA — No formal statistical comparison was conducted; Least-Squares Mean Difference = 0, 95% CI 2-sided [-0.6 to 0.6], Standard Error of Mean 0.3

6. Secondary Outcome: Change in Systolic Blood Pressure (SBP) From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean change in SBP from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin or sitagliptin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 181 | 365 | 360 | 355
mmHg | 1.52 (0.829) | -3.84 (0.602) | -5.06 (0.605) | -1.83 (0.611)
Statistical Analysis 1: Comparison: Placebo/Sitagliptin vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -5.36, 95% CI 2-sided [-7.280 to -3.439], Standard Error of Mean 0.979
Statistical Analysis 2: Comparison: Placebo/Sitagliptin vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -6.58, 95% CI 2-sided [-8.504 to -4.653], Standard Error of Mean 0.981
Statistical Analysis 3: Comparison: Placebo/Sitagliptin vs Sitagliptin 100 mg; Test type: Superiority or Other; ANCOVA — No formal statistical comparison was conducted; Least-Squares Mean Difference = -3.34, 95% CI 2-sided [-5.273 to -1.413], Standard Error of Mean 0.984

7. Secondary Outcome: Percent Change in Triglycerides From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean percent change in triglycerides from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin or sitagliptin group minus placebo) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 171 | 358 | 341 | 338
Percent change | 3.2 (3.6) | 1.6 (2.6) | -1.4 (2.6) | 1.0 (2.7)
Statistical Analysis 1: Comparison: Placebo/Sitagliptin vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.702, ANCOVA; Least-Squares Mean Difference = -1.6, 95% CI [-9.9 to 6.7], Standard Error of Mean 4.2
Statistical Analysis 2: Comparison: Placebo/Sitagliptin vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.274, ANCOVA; Least-Squares Mean Difference = -4.7, 95% CI 2-sided [-13.0 to 3.7], Standard Error of Mean 4.3
Statistical Analysis 3: Comparison: Placebo/Sitagliptin vs Sitagliptin 100 mg; Test type: Superiority or Other; ANCOVA — No formal statistical comparison was conducted; Least-Squares Mean Difference = -2.3, 95% CI 2-sided [-10.6 to 6.1], Standard Error of Mean 4.3

8. Secondary Outcome: Percent Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean percent change in HDL-C from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin or sitagliptin group minus placebo) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 171 | 357 | 336 | 336
Percent change | 3.7 (1.3) | 10.4 (0.9) | 12.1 (1.0) | 5.0 (1.0)
Statistical Analysis 1: Comparison: Placebo/Sitagliptin vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = 6.7, 95% CI 2-sided [3.6 to 9.7], Standard Error of Mean 1.6
Statistical Analysis 2: Comparison: Placebo/Sitagliptin vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = 8.5, 95% CI 2-sided [5.4 to 11.5], Standard Error of Mean 1.6
Statistical Analysis 3: Comparison: Placebo/Sitagliptin vs Sitagliptin 100 mg; Test type: Superiority or Other; ANCOVA — No formal statistical comparison was conducted; Least-Squares Mean Difference = 1.3, 95% CI 2-sided [-1.7 to 4.4], Standard Error of Mean 1.6

9. Secondary Outcome: Change in HbA1c From Baseline to Week 52
Description: The table below shows the least-squares (LS) mean change in HbA1c from Baseline to Week 52 for each active treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus sitagliptin) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 52
Population: Analysis used mITT analysis set (all randomized patients who received at least 1 dose of study drug). Last-observation-carried-forward method used for missing Week 52 values. Measurements taken pre-rescue used as last observation in patients receiving glycemic rescue therapy. Table includes only patients with both baseline and post baseline values.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Canagliflozin 100 mg | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 365 | 360 | 354
Percent | -0.73 (0.047) | -0.88 (0.047) | -0.73 (0.047)
Statistical Analysis 1: Comparison: Canagliflozin 100 mg vs Sitagliptin 100 mg; Test type: Non-Inferiority or Equivalence — Assuming a discontinuation rate of 35% at Week 52, with a 2:2:2:1 treatment assignment ratio for canagliflozin 100 mg, canagliflozin 300 mg, sitagliptin 100 mg, or placebo, it was estimated that 360 subjects would need to be randomly assigned to each of the 3 active treatment groups and approximately 180 subjects to the placebo group to demonstrate non-inferiority with a non-inferiority margin of 0.3%; ANCOVA; Least-Squares Mean Difference = 0.00, 95% CI 2-sided [-0.119 to 0.122], Standard Error of Mean 0.061
Statistical Analysis 2: Comparison: Canagliflozin 300 mg vs Sitagliptin 100 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; ANCOVA; Least-Squares Mean Difference = -0.15, 95% CI 2-sided [-0.273 to -0.031], Standard Error of Mean 0.062

10. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 52
Description: The table below shows the least-squares (LS) mean change in FPG from Baseline to Week 52 for each active treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus sitagliptin) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 52
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Canagliflozin 100 mg | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 365 | 360 | 354
mg/dL | -26.2 (1.814) | -35.2 (1.833) | -17.7 (1.848)
Statistical Analysis 1: Comparison: Canagliflozin 100 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -8.55, 95% CI 2-sided [-13.25 to -3.857], Standard Error of Mean 2.394
Statistical Analysis 2: Comparison: Canagliflozin 300 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -17.5, 95% CI 2-sided [-22.24 to -12.81], Standard Error of Mean 2.404

11. Secondary Outcome: Percent Change in Body Weight From Baseline to Week 52
Description: The table below shows the least-squares (LS) mean percent change in body weight from Baseline to Week 52 for each active treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus sitagliptin) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 52
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Canagliflozin 100 mg | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 365 | 360 | 355
Percent change | -3.8 (0.2) | -4.2 (0.2) | -1.3 (0.2)
Statistical Analysis 1: Comparison: Canagliflozin 100 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -2.4, 95% CI 2-sided [-3.0 to -1.8], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Canagliflozin 300 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -2.9, 95% CI 2-sided [-3.4 to -2.3], Standard Error of Mean 0.3

12. Secondary Outcome: Change in Systolic Blood Pressure (SBP) From Baseline to Week 52
Description: The table below shows the least-squares (LS) mean change in SBP from Baseline to Week 52 for each active treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus sitagliptin) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 52
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Canagliflozin 100 mg | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 365 | 360 | 355
mmHg | -3.53 (0.615) | -4.65 (0.618) | -0.66 (0.625)
Statistical Analysis 1: Comparison: Canagliflozin 100 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -2.87, 95% CI 2-sided [-4.464 to -1.276], Standard Error of Mean 0.812
Statistical Analysis 2: Comparison: Canagliflozin 300 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -3.99, 95% CI 2-sided [-5.589 to -2.389], Standard Error of Mean 0.815

13. Secondary Outcome: Percent Change in Triglycerides From Baseline to Week 52
Description: The table below shows the least-squares (LS) mean percent change in triglycerides from Baseline to Week 52 for each active treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus sitagliptin) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 52
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Canagliflozin 100 mg | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 359 | 343 | 339
Percent change | 1.9 (2.4) | 2.7 (2.4) | -0.4 (2.5)
Statistical Analysis 1: Comparison: Canagliflozin 100 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.466, ANCOVA; Least-Squares Mean Difference = 2.3, 95% CI 2-sided [-3.9 to 8.5], Standard Error of Mean 3.2
Statistical Analysis 2: Comparison: Canagliflozin 300 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.323, ANCOVA; Least-Squares Mean Difference = 3.2, 95% CI 2-sided [-3.1 to 9.4], Standard Error of Mean 3.2

14. Secondary Outcome: Percent Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline to Week 52
Description: The table below shows the least-squares (LS) mean percent change in HDL-C from Baseline to Week 52 for each active treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus sitagliptin) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 52
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Canagliflozin 100 mg | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 359 | 343 | 338
Percent change | 11.2 (1.0) | 13.3 (1.1) | 6.0 (1.1)
Statistical Analysis 1: Comparison: Canagliflozin 100 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = 5.2, 95% CI 2-sided [2.5 to 8.0], Standard Error of Mean 1.4
Statistical Analysis 2: Comparison: Canagliflozin 300 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = 7.3, 95% CI 2-sided [4.5 to 10.1], Standard Error of Mean 1.4

ADVERSE EVENTS:
Time Frame: Adverse events were reported for the duration of the study; each patient participated in the study for approximately 52 weeks.
Description: The total number of adverse events listed in the "Other (non-Serious) Adverse Event" table are based upon a cut-off of greater than or equal to 5 percent of patients experiencing the adverse event in any treatment arm.
Groups:
- Placebo/Sitagliptin: Baseline to Week 26: Each patient received matching placebo once daily for 26 weeks and were then switched from placebo to 100 mg of sitagliptin once daily until Week 52. Placebo and sitagliptin were given with protocol-specified doses of metformin immediate release. Data are presented for Baseline to Week 26.
- Canagliflozin 100 mg: Baseline to Week 26: Each patient received 100 mg of canagliflozin once daily for 52 weeks with protocol-specified doses of metformin immediate release. Data are presented for Baseline to Week 26.
- Canagliflozin 300 mg: Baseline to Week 26: Each patient received 300 mg of canagliflozin once daily for 52 weeks with protocol-specified doses of metformin immediate release. Data are presented for Baseline to Week 26.
- Sitagliptin 100 mg: Baseline to Week 26: Each patient received 100 mg of sitagliptin once daily for 52 weeks with protocol-specified doses of metformin immediate release. Data are presented for Baseline to Week 26.
- Placebo/Sitagliptin: Baseline to Week 52: Each patient received matching placebo once daily for 26 weeks and were then switched from placebo to 100 mg of sitagliptin once daily until Week 52. Placebo and sitagliptin were given with protocol-specified doses of metformin immediate release. Data are presented for Baseline to Week 52.
- Canagliflozin 100 mg: Baseline to Week 52: Each patient received 100 mg of canagliflozin once daily for 52 weeks with protocol-specified doses of metformin immediate release. Data are presented for Baseline to Week 52.
- Canagliflozin 300 mg: Baseline to Week 52: Each patient received 300 mg of canagliflozin once daily for 52 weeks with protocol-specified doses of metformin immediate release. Data are presented for Baseline to Week 52.
- Sitagliptin 100mg: Baseline to Week 52: Each patient received 100 mg of sitagliptin once daily for 52 weeks with protocol-specified doses of metformin immediate release. Data are presented for Baseline to Week 52.
Arm/Group | Placebo/Sitagliptin: Baseline to Week 26 | Canagliflozin 100 mg: Baseline to Week 26 | Canagliflozin 300 mg: Baseline to Week 26 | Sitagliptin 100 mg: Baseline to Week 26 | Placebo/Sitagliptin: Baseline to Week 52 | Canagliflozin 100 mg: Baseline to Week 52 | Canagliflozin 300 mg: Baseline to Week 52 | Sitagliptin 100mg: Baseline to Week 52
Serious Adverse Events (participants affected / at risk) | 4/183 | 12/368 | 10/367 | 8/366 | 7/183 | 15/368 | 12/367 | 18/366
Other Adverse Events (participants affected / at risk) | 31/183 | 55/368 | 45/367 | 42/366 | 55/183 | 108/368 | 101/367 | 109/366
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Sitagliptin: Baseline to Week 26 (N=183) | Canagliflozin 100 mg: Baseline to Week 26 (N=368) | Canagliflozin 300 mg: Baseline to Week 26 (N=367) | Sitagliptin 100 mg: Baseline to Week 26 (N=366) | Placebo/Sitagliptin: Baseline to Week 52 (N=183) | Canagliflozin 100 mg: Baseline to Week 52 (N=368) | Canagliflozin 300 mg: Baseline to Week 52 (N=367) | Sitagliptin 100mg: Baseline to Week 52 (N=366)
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Cataract nuclear (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52. NOTE: event was reassessed as non-serious in the Week 52 study report.
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52. In the Week 26 study report, this event was coded as "abdominal pain"; it was subsequently re-coded in the Week 52 study report as "abdominal hernia".
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Hernia obstructive (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52. In the Week 26 study report, this event was coded as "hernia obstructive"; it was subsequently re-coded in the Week 52 study report as "incisional hernia, obstructive".
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Pyothorax (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52. In the Week 26 study report, this event was coded as "pyothorax"; it was subsequently re-coded in the Week 52 study report as "infectious pleural effusion".
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Malignant mesenchymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Coma (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
High risk pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Arterial thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52. In the Week 26 study report, this event was coded as "abdominal pain"; it was subsequently re-coded in the Week 52 study report as "abdominal hernia".
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52. In the Week 26 study report, this event was coded as "pyothorax"; it was subsequently re-coded in the Week 52 study report as "infectious pleural effusion".
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52. In the Week 26 study report, this event was coded as "hernia obstructive"; it was subsequently re-coded in the Week 52 study report as "incisional hernia, obstructive".
Multiple drug overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Large cell lung cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Sitagliptin: Baseline to Week 26 (N=183) | Canagliflozin 100 mg: Baseline to Week 26 (N=368) | Canagliflozin 300 mg: Baseline to Week 26 (N=367) | Sitagliptin 100 mg: Baseline to Week 26 (N=366) | Placebo/Sitagliptin: Baseline to Week 52 (N=183) | Canagliflozin 100 mg: Baseline to Week 52 (N=368) | Canagliflozin 300 mg: Baseline to Week 52 (N=367) | Sitagliptin 100mg: Baseline to Week 52 (N=366)
Diarrhoea (Gastrointestinal disorders) | 12 | 12 | 18 | 16 | 13 | 15 | 23 | 23 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Nasopharyngitis (Infections and infestations) | 13 | 15 | 10 | 14 | 13 | 18 | 16 | 22 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Headache (Nervous system disorders) | 12 | 12 | 10 | 16 | 13 | 19 | 13 | 19 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Pollakiuria (Renal and urinary disorders) | 1 | 21 | 10 | 2 | 1 | 21 | 11 | 2 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Upper respiratory tract infection (Infections and infestations) | 6 | 5 | 18 | 18 | 10 | 12 | 23 | 22 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Urinary tract infection (Infections and infestations) | 4 | 18 | 13 | 12 | 12 | 27 | 17 | 22 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 7 | 4 | 11 | 11 | 10 | 9 | 17 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 8 | 12 | 4 | 10 | 13 | 15 | 10 — Source vocabulary is MEDDRA 14.0 for Week 26 and MEDDRA 15.0 for Week 52.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.